CLINICAL TRIAL: NCT00171964
Title: Evaluation of the Efficacy and Tolerability of Zoledronic Acid in Combination With Radiotherapy in Patients With Advanced Osteolytic Bone Lesions
Brief Title: Efficacy and Tolerability of Zoledronic Acid With Radiotherapy in Pts With Advanced Osteolytic Bone Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EDE06
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2012-04

CONDITIONS: Pain; Neoplasm Metastasis; Cancer
Keywords: Pain; Bone metastasis; Analgesic consumption; Cancer patients; Cancer patients with painful bone metastasis
MeSH Terms: conditions — Pain; Neoplasm Metastasis; Neoplasms | interventions — Zoledronic Acid; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- zoledronic acid + radiotherapy (Experimental): zoledronic acid every 4 weeks in combination with radiotherapy
  Interventions: Drug: Zoledronic acid in combination with therapy

INTERVENTIONS:
Drug: Zoledronic acid in combination with therapy
  Other Names: Zometa; Zomera; Aclasta; Reclast

SUMMARY:
It is the aim of this multicentric clinical study to assess the efficacy and tolerability of zoledronic acid in combination with radiotherapy in patients with advanced osteolytic bone lesions in terms of the reduction of pain and analgesic consumption.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least one cancer-related bone lesion in cancer patients, confirmed by X-ray, MRT or computer tomography
* Severity of pain ≥ 5 on item 3 of the BPI which is caused by the bone lesion(s) and requires radiotherapy
* Adequate liver function - serum total bilirubin concentration less than 1.5 x the upper limit of normal value
* Expected survival time ≥ 6 months
* If the patient is of child-bearing potential: negative pregnancy test at screening
* ECOG performance status of 0, 1 or 2.
* Written informed consent

Exclusion Criteria:

* Prior treatment with an oral bisphosphonate for more than 3 months or more than 3 intravenous (i.v.) bisphosphonate applications
* Bisphosphonate treatment within 6 months before study start
* Previous radiotherapy of the painful areas to be irradiated. An initiation of radiotherapy for the target area(s) up to 3 days at maximum prior to the first infusion is allowed.
* Skeleton-related complications (e.g., pathological fractures, orthopedic intervention to treat or stabilize an osteolytic defect, spinal cord compression) during the last 3 weeks prior to the first infusion of trial medication.
* Initiation of a new chemotherapeutic treatment regimen during the last 2 weeks prior to the first infusion of trial medication
* Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute. Creatinine clearance (CrCl) is calculated using the Cockcroft-Gault formula: CrCl = [140-age (years)] x weight (kg) {x 0.85 for female patients} [72 x serum creatinine (mg/dL)]
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or ≥ 12.0 mg/dl (3.00 mmol/L).
* Patients with clinically symptomatic brain metastases
* History of diseases with influence on bone metabolism such as Paget's disease and primary hyperparathyroidism
* Pregnancy and lactation
* Women of childbearing potential not on a medically recognized form of contraception (i.e., oral contraceptives or implants, intrauterine device [IUD], vaginal diaphragm or sponge, or condom with spermicide)
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction | weekly assessments during 48 weeks

SECONDARY OUTCOMES:
Time to pain reduction | weeks 0, 12, 24, 36, 48 and 60
Duration of pain reduction | weeks 0, 12, 24, 36, 48 and 60
Quality of life | weeks 0, 12, 24, 36, 48 and 60
Changes in parameters of bone turnover | weeks 0, 12, 24, 36, 48 and 60

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Herne, Germany

REFERENCES:
- See also: Related Info — http://link.springer.com/article/10.1007/s00066-011-1001-z